CLINICAL TRIAL: NCT05954676
Title: Effects of Online Peri-operative Education Program for Patients Undergoing Major Head & Neck Surgery
Brief Title: Online Peri-operative Education Program for Patients Undergoing Major Head & Neck Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Zero accruals
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201909127
Record Dates: First submitted 2023-07-10; First posted 2023-07-20 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer; Head and Neck Neoplasms
Keywords: Head and neck cancer; CareOrbit; Peri-operative education
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CareOrbit - Patients (Experimental): Patients will be assigned a username and password to access their CareOrbit account via the internet (caregivers will use the same account information). These patients may designate up to 3 additional individuals who will be participating in the patient's postoperative care to receive the link along with a unique username and password via email. All patients will additionally receive standard pre- and post-operative instructions and care. This will include verbal education by the surgeons at their pre-operative visits.
  Patient questionnaires will be distributed at the first and second post-operative visits (typically 1-2 weeks after discharge and 3 months after post-operative clinic visit). At 30 days following discharge, the patients' medical records will be reviewed by the study team to assess for the primary or secondary outcomes. Patients will be contacted by telephone to inquire about ED/UC visits outside of the BJC system.
  Interventions: Other: CareOrbit
- CareOrbit - Caregivers (Experimental): Patients will be assigned a username and password to access their CareOrbit account via the internet (caregivers will use the same account information). These patients may designate up to 3 additional individuals who will be participating in the patient's postoperative care to receive the link along with a unique username and password via email. All patients will additionally receive standard pre- and post-operative instructions and care. This will include verbal education by the surgeons at their pre-operative visits.
  Patient questionnaires will be distributed at the first and second post-operative visits (typically 1-2 weeks after discharge and 3 months after post-operative clinic visit). At 30 days following discharge, the patients' medical records will be reviewed by the study team to assess for the primary or secondary outcomes. Patients will be contacted by telephone to inquire about ED/UC visits outside of the BJC system.
  Interventions: Other: CareOrbit

INTERVENTIONS:
Other: CareOrbit — CareOrbit is a third-party organization that provides a HIPAA-compliant, patient-centered digital engagement platform that helps create, organize, and update content to educate and serve the patient and caregivers through their entire treatment journey.

SUMMARY:
This phase of the project will evaluate the utility and efficacy of a personalized online patient education platform developed from efforts in Phase 1 in 1) increasing patients' and caregivers' pre- and post-operative preparedness and satisfaction, and 2) reducing readmission, ED/Urgent care/unplanned clinic visits and telephone calls to clinic staff.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have had or are undergoing free flap surgery and/or total laryngetomy
* Have internet access
* English speaking

Exclusion Criteria:

* Younger than 18 years of age
* No internet access
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
30-day readmission | At Day 30

SECONDARY OUTCOMES:
Number of emergency room/urgent care visits | Through 3 months post-operative
Number of unplanned clinic visits | Through 3 months post-operative
Number of telephone calls/electronic messages to clinic staff | Through 3 months post-operative
Satisfaction of education | At pre-operative visit, 2 weeks post-operative, and 3 months post-operative
  Participants will complete a survey asking satisfaction of the educational material. Answers range from 1=excellent to 5=poor. A higher score indicates a higher level of satisfaction.
Preparedness for head and neck surgery and post-operative care | At pre-operative visit, 2 weeks post-operative, and 3 months post-operative
  Participants will complete a survey asking satisfaction of the educational material. Answers range from 1=excellent to 5=poor. A higher score indicates a higher level of preparedness.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Rich, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No